CLINICAL TRIAL: NCT01530555
Title: Prospective Phase II Study of Rabbit Antithymocyte Globulin (ATG, Thymoglobuline®, Genzyme) With Ciclosporin for Patients With Acquired Aplastic Anaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2081-005
Record Dates: First submitted 2012-01-24; First posted 2012-02-10 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-02

CONDITIONS: Acquired Aplastic Anaemia
MeSH Terms: interventions — thymoglobulin; Antilymphocyte Serum

ARMS (1):
- Treatment arm (Experimental): 1. Rabbit ATG, Thymoglobuline (Genzyme) 1.5 vials/10kg (3.75mg/kg) daily for 5 days given as an intravenous infusion over 12-18 hours.
  2. Ciclosporin (CSA) 5mg/kg/day orally from day +1 for a minimum of 6 months, with later tailing according to individual patient response. Aim to maintain trough whole blood CSA levels between 150 and 250 ng/ml.
  Interventions: Drug: Rabbit ATG, Thymoglobuline (Genzyme)

INTERVENTIONS:
Drug: Rabbit ATG, Thymoglobuline (Genzyme) — 1. Rabbit ATG, Thymoglobuline® (Genzyme) 1.5 vials/10kg (3.75mg/kg) daily for 5 days given as an intravenous infusion over 12-18 hours.
  2. Ciclosporin (CSA) 5mg/kg/day orally from day +1 for a minimum of 6 months

SUMMARY:
To assess the tolerability and efficacy of rabbit antithymocyte globulin (ATG, Thymoglobuline®) with ciclosporin (CSA) in the first line treatment of patients with acquired severe aplastic anaemia (SAA), and patients with non-severe aplastic anaemia (NSAA) and who are transfusion dependent. To compare the response rate of the combination of rabbit ATG (Thymoglobuline® and CSA from this pilot study with the response rate observed in a series of matched AA patients; treated after 1994 with the combination of horse ATG (Lymphoglobuline®) and CSA; obtained from the EBMT database (comparative study).

ELIGIBILITY:
Inclusion Criteria:

1. To define aplastic anaemia there must be at least two of the following: (1) haemoglobin < 10g/dl; (2) platelet count < 50 x 109/l; (3) neutrophil count < 1.5 x 109/l, and a hypocellular bone marrow on bone marrow biopsy
2. Time from diagnosis to study registration ≤ 6mths
3. No prior treatment except for haemopoietic growth factors given for no more than 4 weeks, and androgens.
4. Age ≥ 16yrs (≥ 18yrs in Germany in accordance with German law), with no upper age limit.

Exclusion criteria:

1. Eligibility for an HLA-matched sibling donor transplant for SAA patients
2. Prior therapy with ATG or CSA
3. Haematopoeitic growth factors more than 4 weeks before study enrollment
4. Diagnosis of Fanconi anaemia, dyskeratosis congenita or congenital bone marrow failure syndrome
5. Evidence of myelodysplastic disease
6. Paroxysmal nocturnal haemoglobinuria with evidence of significant haemolysis, history of PNH associated thrombosis or a PNH clone > 50% by flow cytometry
7. Diagnosis or previous history of carcinoma (except local cervical, basal cell, squamous cells, or melanoma)
8. Subject is pregnant (e.g. positive HCG test) or is breast feeding
9. Severe uncontrolled infection or unexplained fever > 38oC
10. Subjects who have hepatic, renal cardiac, metabolic or other concurrent diseases of such severity that life expectancy is less than 3 months

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Response | 2 years
  Primary outcome is response at 6 months post ATG treatment

SECONDARY OUTCOMES:
Over all survival | 2 years
  Secondary outcome variables include overall survival and failure free survival at 2 years post ATG treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Al Zahrani, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center